CLINICAL TRIAL: NCT04227418
Title: An Evaluation of the Safety and Clinical Utility of Handheld ECG Technology in Psychiatry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: Leeds and York Partnership NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: EVALECG MEPS Study
Record Dates: First submitted 2019-11-04; First posted 2020-01-13 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular Diseases; Dementia; Mental Health Disorder
MeSH Terms: conditions — Cardiovascular Diseases; Dementia; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mental Health
  Interventions: Device: 12 lead ECG monitoring; Device: 6 lead ECG monitoring; Device: Hand held ECG monitoring
- Psychiatric
  Interventions: Device: 12 lead ECG monitoring; Device: 6 lead ECG monitoring; Device: Hand held ECG monitoring

INTERVENTIONS:
Device: 12 lead ECG monitoring — Rate, Rhythm, QTc and PR interval will be assessed
Device: 6 lead ECG monitoring — Rate, Rhythm, QTc and PR interval will be assessed
Device: Hand held ECG monitoring — Handheld ECG machines are portable, inexpensive, hand held devices that provide a 'real-time' rhythm strip, equivalent to lead I or II on a 12 lead machine, depending on how the device is held. The rhythm strip is displayed on a computer tablet or mobile phone, and are compatible with both android and iPhone platforms. To perform the test the patient places their fingers/thigh, or alternatively the device can be placed directly on the patient's chest. The process does not require the patient to be exposed, can be done in a seated position (negating the need an examination couch) and their ease of use and portability means they could be readily used in memory clinics or community settings.
  Other Names: AliveCor ECG device

SUMMARY:
Acetylcholinesterase inhibitors and antipsychotics are drugs commonly prescribed in psychiatry, the former for dementia and the latter for acute and chronic psychotic illness. Both can cause cardiac arrhythmia therefore 12 lead ECG's are recommended before prescribing. The test is often difficult to obtain however, leading to either patients being inconvenienced or drugs prescribed without the test. There are two parts of this study, but both examine the utility of single lead ecg monitoring, one in the memory clinic and the other in inpatient psychiatry wards. The aim to to evaluate the safety and efficacy of the handheld ecg versus the 12 lead and 6 lead ecg, and whether the handheld ecg can be used to screen for ecg abnormalities that would generally lead to a caution or contra-indication for acetylcholinesterase inhibitors and anti-psychotic medication.

Patients will either be recruited from the outpatient memory clinic or in patient psychiatry wards. Following informed consent baseline demographic data will be collected, and patients will undergo a 12 lead and 6 lead ECG as well as a rhythm strip using the handheld device. Data from this point will be annonymised for future analysis. The psychiatrists ECG report will also be recorded, and a subset of patients will undergo an echocardiogram (to see what proportion of patients with psychiatric disorders have structural heart disease.)

ELIGIBILITY:
Inclusion Criteria:

Any patient attending the memory clinic Any patient admitted to the acute psychiatric ward requiring antipsychotic medication

Exclusion Criteria:

Patients who lack capacity and do not have a personal consultee to provide assent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults, 18 and over, attending memory clinic with a new diagnosis of Alzheimer's, Mixed or Lewy Body type dementia indicated for AChIE treatment, will be invited to participate. These are patients who would be indicated to have an ECG as part of routine practice.
  All general adult and old age inpatient wards in Leeds and York Partnership NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
ECG monitoring | 45 minutes
  12 lead, 6 lead and handheld ECG device monitoring will be undertaken.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Partnership NHS Foundation Trust, Leeds, West Yorkshire, United Kingdom